CLINICAL TRIAL: NCT06914076
Title: Evaluating The Effectiveness Of Structured Psychosocial Counseling On Mental Health And Functional Independence In Individuals With Low Vision
Brief Title: Evaluating The Effectiveness Of Structured Psychosocial Counseling On Mental Health And FI Individuals With Low Vision
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/814
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Psychosocial Counseling (Experimental)
  Interventions: Combination Product: Structured Psychosocial Counseling
- Standard Care (Active Comparator)
  Interventions: Diagnostic Test: Standard Care

INTERVENTIONS:
Combination Product: Structured Psychosocial Counseling — "Group A (Experimental Group):
  Participants in the Experimental group will be divided into groups with the persons having visual acuity 6/60, counting fingers and light perception will receive low vision aids etc and structured psychosocial counseling tailored for individuals with low vision. Counseling will be delivered over a 12-week period, consisting of weekly 60-minute sessions conducted by trained counselors. The program will focus on the following:
  Coping mechanisms for depression and anxiety. Strategies to improve functional independence and daily living skills. Social integration techniques to enhance participation in community activities. Low visions aids under supervision of low vision specialist."
  Arms: Structured Psychosocial Counseling
Diagnostic Test: Standard Care — Group B (Control Group): The control group will continue receiving standard care, including referrals and informational support.
  Arms: Standard Care

SUMMARY:
Vision impairments affect 2.2 billion people worldwide, including 36 million who are blind and 217 million with moderate-to-severe visual impairment. In the US, age-related vision loss is a leading cause of disability among older adults.

DETAILED DESCRIPTION:
With increasing longevity, global blindness rates are expected to triple, and moderate-to-severe vision impairment rates to double in 30 years. The study aims to assess the effects of structured psychosocial counseling on mental health (depression, anxiety) and functional independence in individuals with low vision. Additionally, it seeks to evaluate the overall impact on quality of life (QoL) following the counseling intervention. A randomized controlled trial will be conducted at Superior University Lahore.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 80 years.
* Both male and female
* Individuals diagnosed with low vision, defined as a visual acuity of less than 6/18 but equal to or better than 3/60 in the better eye with best correction.
* Individuals having visual acuity 6/60, Counting fingers or light perception.
* Individuals experiencing symptoms of depression or anxiety as assessed through a validated screening tool.
* Individuals reporting reduced functional independence in daily activities due to low vision.

Exclusion Criteria:

* Unable to provide informed consent.
* Diagnosed with severe psychiatric disorders such as schizophrenia, bipolar disorder, or severe post-traumatic stress disorder.
* Existing involvement in similar counseling programs.
* Presence of medical conditions or disabilities.
* Pregnant individuals if pregnancy-related complications or responsibilities could interfere with participation in the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
DASS 21 | 12 Months
  The DASS-21 uses the following categories to interpret scores:
  Normal: 0-9 (Depression), 0-7 (Anxiety), 0-14 (Stress) Mild: 10-13 (Depression), 8-9 (Anxiety), 15-18 (Stress) Moderate: 14-20 (Depression), 10-14 (Anxiety), 19-25 (Stress) Severe: 21-27 (Depression), 15-19 (Anxiety), 26-33 (Stress) Extremely Severe: 28+ (Depression), 20+ (Anxiety), 34+ (Stress)
LVQoL Questionare | 12 Months
  Total Score Interpretation:
  * 25-50: Good quality of life
  * 51-75: Moderate quality of life
  * 76-100: Poor quality of life
  * 101-125: Very poor quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Dial hospital, Qadirabad road Ali pur chattah, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No